CLINICAL TRIAL: NCT00620191
Title: Metformin in the Prevention of Alzheimer's Disease
Brief Title: Metformin in Amnestic Mild Cognitive Impairment
Acronym: MCI
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Columbia University (Other)
Collaborators: Institute for the Study of Aging (ISOA) (Other); National Institute on Aging (NIA) (NIH)
Responsible Party: Principal Investigator, José A. Luchsinger, Associate Professor of Medicine and Epidemiology at NYPH/CUMC, Columbia University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: AAAC7231; R01AG026413 (NIH); 270901 (Other Grant/Funding Number: Alzheimer's Disease Drug Discovery Foundation)
Record Dates: First submitted 2008-02-07; First posted 2008-02-21 (Estimated); Results first posted 2020-10-23 (Actual); Last update posted 2020-10-23 (Actual); Status verified 2020-09

CONDITIONS: Mild Cognitive Impairment
Keywords: Metformin; Mild Cognitive Impairment (MCI); Alzheimer's Disease (AD); Overweight; Insulin
MeSH Terms: conditions — Cognitive Dysfunction; Alzheimer Disease; Overweight; Insulin Resistance | interventions — Metformin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Matching Placebo (Placebo Comparator): Placebo identical to metformin
  Interventions: Drug: Placebo
- Metformin (Experimental): Metformin 1000 mg twice a day
  Interventions: Drug: Metformin

INTERVENTIONS:
Drug: Metformin — Metformin 1000 mg twice a day titrated from 500 mg once a day
  Other Names: Glucophage
  Arms: Metformin
Drug: Placebo — Placebo identical to metformin 2 tablets twice a day titrated from one table once a day
  Arms: Matching Placebo

SUMMARY:
Hyperinsulinemia and type 2 diabetes (T2D) are important potential risk factors for cognitive decline and Alzheimer's disease (AD). Two thirds of the US adult population are at risk for hyperinsulinemia and T2D, and half of the population 85 years and older have AD. Peripheral hyperinsulinemia can impair the clearance of amyloid beta in the brain, the main culprit in AD. Thus, the investigators hypothesize that lowering peripheral insulin in overweight persons with amnestic mild cognitive impairment (AMCI), a transition state between normal cognition and AD, can decrease the risk of cognitive decline and progression to AD. The investigators propose to conduct a phase II double blinded placebo controlled randomized clinical trial of metformin, a safe and effective medication that prevents hyperinsulinemia and diabetes, to test this hypothesis among 80 overweight persons aged 55 to 90 years with AMCI. The main outcome of the study will be changes in performance in a memory test (total recall of the Selective Reminding Test) and the Score a test of general cognitive function used in clinical trials (the Alzheimer's Disease Assessment Scale-cognitive subscale (ADAS-Cog)). Another aim is to compare brain function in an area affected by Alzheimer's disease between the metformin and placebo group mean changes from beginning to end among 40 participants using a PET scan.

DETAILED DESCRIPTION:
The prevalence of Alzheimer's disease (AD) is expected to quadruple by the year 2047. There are no known curative or preventive measures for AD. Current treatment options for AD only address symptoms, and no treatments are available that focus on delaying the actual disease process. One of the currently accepted hypothesis of the pathogenesis of AD is that the main culprit is the accumulation of Aβ in the brain, and this process has become a target for treatments and preventive measures. Amnestic mild cognitive impairment (MCI) has been used to describe a transitional state between normal cognitive function and AD, and has thus been targeted for interventions. Persons with MCI progress to AD at the rate of nearly 10% to 15% per year. The criteria most commonly used for the definition of AD dementia from MCI. The investigators propose to use these criteria with slight modification to recruit persons for a pilot trail of AD prevention in persons with amnestic MCI.

Peripheral hyperinsulinemia (high insulin levels) potentially impair Aβ clearance, and in this study we are proposing to use metformin, an insulin lowering agent, to prevent AD by improving Aβ clearance in the brain. The insulin resistance syndrome and hyperinsulinemia are common in individuals with and without diabetes, and are related to increased risk of cardiovascular and cerebrovascular outcomes. Hyperinsulinemia predicts the development of diabetes; therefore, diabetes can be considered a consequence and a marker of past hyperinsulinemia. According to NHANES III data, more than 40% of the population over the age of 60 years has problems of glucose intolerance or diabetes, all related to insulin resistance and hyperinsulinemia. The investigators have found that the risk of AD in individuals without diabetes increases with increasing levels of fasting insulin, and that high insulin levels are related to a faster decline in memory scores. The high prevalence of hyperinsulinemia and diabetes (49% of the elderly in Northern Manhattan) and its biological plausibility as a risk factor for cognitive decline and AD has attracted increasing attention. In this application we are targeting hyperinsulinemia, the most important risk factor for AD identified in the elderly population of Northern Manhattan. The risk of AD attributable to hyperinsulinemia or diabetes in Northern Manhattan was 39%, and is higher in Hispanics and African-Americans, who have a higher prevalence of diabetes and insulin resistance, and will comprise the majority of our sample.

ELIGIBILITY:
Inclusion criteria:

* Age range: 55 years to 90 years. The main rationale for this inclusion criteria is to follow the standard set by the Alzheimer's Disease Cooperative Study (ADCS).
* Memory complaint expressed by the participant and recognized by the informant. The memory complaint must represent a change from previous functioning based on information provided by both subject and informant.
* Fluent in English or Spanish.
* Mini-Mental State Examination (MMSE) equal or more than 20.
* Subjects must fulfill criteria for amnestic mild cognitive impairment (MCI). Guidelines for the diagnosis of MCI: Subjects must score below a predetermined cut-off score on the logical memory II delayed paragraph recall sub-test of the Wechsler Memory Scale Revised (WMS-R) or the selective reminding test (SRT).
* Global Clinical Dementia Rating (CDR) score must be 0.5 at screening.
* Subjects without a known history of diabetes or diabetes that has never been treated with medications. If diabetes is diagnosed during screening or they have a history of diabetes not treated in the last 12 months they will be excluded if their Hemoglobin A1c (HbA1c) is > 6.5. In addition, a diagnosis of diabetes can be made if the HbA1c is 6.5% or more.
* Overweight or obese by National Heart, Lung, and Blood Institute (NHLBI) criteria (Body Mass Index (BMI) of more or equal of 25 kg/ m2).
* No contraindications to metformin treatment.
* Hachinski score less or equal to 4.
* Hamilton score less or equal to 12 on the 17 item scale.
* General cognition and functional performance such that a diagnosis of dementia cannot be made at the time of screening based on DSM-IV criteria.
* Vision and hearing must be sufficient for compliance with testing procedures.

Exclusion criteria:

* Individuals with dementia
* MMSE < 20
* Subjects with neurologic diseases associated to neurologic deficits.
* Subjects with current psychiatric diagnoses such as depression, bipolar disorder or schizophrenia.
* Subjects with uncontrolled hypertension (systolic blood pressure more than 160 mmHg or diastolic blood pressure more than 95 mmHg.
* Subjects with a history of active cancer or cancer within last five years, with the exception of squamous or basal cell carcinoma of the skin.
* Subjects who for any reason may not complete the study as judged by the study physician.
* Subjects with a known history of diabetes treated with medications.
* Subjects with a new or old diagnosis of diabetes, never treated, with a HbA1c of more than 6.5 .
* Contraindications to metformin: Contraindications to metformin use include a creatinine of > 1.5, liver disease by history or by elevated transaminases, congestive heart failure, and alcohol abuse.
* Use of cholinesterase inhibitors.

Exclusion criteria for brain imaging study:

* Presence of diabetes, even if the HbA1c is less or equal to 6.5.
* Inability to lie down for any reason.
* Presence of any metallic implant.
* Claustrophobia.
* Any contraindication to magnetic resonance imaging (MRI) or fluorodeoxyglucose (FDG) positron emission tomography (PET).

Ages: 55 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2008-06-01 (Actual); Primary Completion 2012-02 (Actual); Study Completion 2012-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jose A Luchsinger, MD, Principal Investigator — Columbia University
Locations (1):
- Columbia University Medical Center, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Luchsinger JA, Perez T, Chang H, Mehta P, Steffener J, Pradabhan G, Ichise M, Manly J, Devanand DP, Bagiella E. Metformin in Amnestic Mild Cognitive Impairment: Results of a Pilot Randomized Placebo Controlled Clinical Trial. J Alzheimers Dis. 2016;51(2):501-14. doi: 10.3233/JAD-150493. PMID 26890736

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment was completed in 32 months (2.5 subjects a month) [38]; 1426 subjects were screened by telephone and 331 were screened in person.
Pre-assignment Details: 1426 screened by telephone and 1095 excluded; 331 deemed eligible for in-person screen; 224 of those were excluded; 87 met eligibility criteria, 7 declined randomization, 80 were randomized
Groups:
- Placebo: placebo identical to metformin.
  placebo: placebo identical to metformin 2 tablets twice a day titrated from one table once a day
Period: Overall Study
Arm/Group | Placebo | Metformin
Started | 40 | 40
3 Month Follow-up | 39 | 39
6 Month Follow-up | 38 | 36
9 Month Follow-up | 37 | 34
Completed | 33 (12 month follow-up) | 32 (12 month follow-up)
Not Completed | 7 | 8

BASELINE CHARACTERISTICS:
Groups:
- Placebo: placebo identical to metformin.
  placebo: placebo identical to metformin 2 tablets twice a day titrated from one table once a day. Participants remained on the maximum number of tolerated tablets (0,1,2,3,4).
- Metformin: metformin 1000 mg twice a day
  metformin: metformin 1000 mg twice a day titrated from 500 mg once a day.Participants remained on the maximum number of tolerated tablets (0,1,2,3,4).
- Total: Total of all reporting groups
Arm/Group | Placebo | Metformin | Total
Number analyzed (Participants) | 40 | 40 | 80
Age, Continuous [Mean (Standard Deviation); unit: Years] | 64.1 (7.9) | 65.3 (7.0) | 64.5 (7.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 24 | 18 | 42
  Male | 16 | 22 | 38
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 13 | 17 | 30
  Not Hispanic or Latino | 27 | 23 | 50
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 15 | 11 | 26
  White | 12 | 12 | 24
  More than one race | 13 | 17 | 30
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 40 | 40 | 80
APOE Epsilon 4 [Number; unit: participants] — homozygous or heterozygous for APOE Epsilon 4
  participants
    ApoE Epsilon 4 positive | 11 | 10 | 21
    ApoE epsilon 4 negative | 29 | 30 | 59
Body Mass Index [Mean (Standard Deviation); unit: kg/m⌃2] | 31.3 (4.7) | 30.9 (4.1) | 31.1 (4.4)
Hemoglobin A1c [Mean (Standard Deviation); unit: percent HbA1c] | 6.1 (0.5) | 6.1 (0.8) | 6.1 (0.6)
Fasting insulin [Mean (Standard Deviation); unit: IU/dl] | 13.4 (7.6) | 16.3 (9.5) | 14.7 (8.6)
Systolic blood pressure [Mean (Standard Deviation); unit: mmHg] | 132.1 (12.4) | 130.8 (10.9) | 131.4 (11.6)
Total Cholesterol [Mean (Standard Deviation); unit: mg/dl] | 208.2 (46.7) | 204.2 (43.6) | 206.2 (44.9)
High Density lipoprotein [Mean (Standard Deviation); unit: mg/dl] | 58.3 (17.7) | 51.5 (14.1) | 54.8 (16.2)
Score of the Alzheimer's Disease Assessment Scale-cognitive subscale (ADAS-cog) [Mean (Standard Deviation); unit: score] — The ADAS-cog is an aggregate for several cognitive tests intended to provide a global cognitive score and consists of 11 tasks. The tasks (and corresponding score range)) are Word Recall (0-10), Naming (0-4), Commands (0-5), Constructional Praxis (0-5) Ideational Praxis (0-5), Orientation (0-8), Word Recognition (0-12), Language (0-5), Word Finding Difficulty (0-5), and Remembering Test Instructions (1-5). The range of aggregate scores (sum of scores) is 1 to 69, with higher scores meaning worse cognitive performance.
  score | 14.6 (6.1) | 12.0 (4.0) | 13.3 (5.3)
Selective Reminding Test Total Recall score [Mean (Standard Deviation); unit: score] — The Selective Reminding Test measures verbal learning and delayed recall through a multiple-trial list-learning paradigm. Patients are presented aurally with a list of 12 words for trial 1 and are asked to recall as many as possible. For trials 2-6, there is a selective presentation of only those words not recalled on the previous trial. Trial 7 is similar to the other trials but is assessed after an 11-minute delay. The score for the selective reminding test is the unweighted average of seven individual study results (min=0 and max=84) Higher scores indicate a better cognitive performance.
  score | 36.1 (9.5) | 34.2 (7.9) | 35.2 (8.7)
Education in Years [Mean (Standard Deviation); unit: Years] | 13.1 (4.5) | 13.8 (3.4) | 13.4 (4.0)

OUTCOME MEASURES:

1. Primary Outcome: Change in Total Recall Score in the Selective Reminding Test
Description: The Selective Reminding Test measures verbal learning and delayed recall through a multiple-trial list-learning paradigm. Patients are presented aurally with a list of 12 words for trial 1 and are asked to recall as many as possible. For trials 2-6, there is a selective presentation of only those words not recalled on the previous trial. Trial 7 is similar to the other trials but is assessed after an 11-minute delay. The score for the selective reminding test is the unweighted average of seven individual study results (min=0 and max=84) Higher scores indicate a better cognitive performance. The total recall score from the first visit was subtracted from that of the last visit to calculate the change in score (total words recalled).
Time Frame: 12 months
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- Placebo: Placebo identical to metformin.
  placebo: placebo identical to metformin 2 tablets twice a day titrated from one tablet once a day. Participants remained on the highest tolerated dose (0,1,2,3,4 tablets).
- Metformin: Metformin 1000 mg twice a day
  metformin: metformin 1000 mg twice a day titrated from 500 mg once a day. Participants remained on the highest tolerated dose (0,1,2,3,4 tablets of 500 mg each).
Arm/Group | Placebo | Metformin
Number analyzed (Participants) | 40 | 40
score on a scale | 5.7 (8.7) | 9.4 (8.5)
Statistical Analysis 1: Comparison: Placebo vs Metformin; Test type: Superiority or Other; p = 0.05, t-test, 2 sided; Mean Difference (Net) = 3.7, Standard Deviation 1.92 — The difference is the value for the metformin arm minus the value for the placebo arm
Statistical Analysis 2: Comparison: Placebo vs Metformin; Test type: Superiority or Other; p = 0.05, ANCOVA; adjusted for baseline ADAS-Cog value; Mean Difference (Net) = 4.1, Standard Deviation 1.36 — The difference is the value for the metformin arm minus the value for the placebo arm

2. Primary Outcome: Change in Score of the Alzheimer's Disease Assessment Scale-cognitive Subscale (ADAS-cog)
Description: The ADAS-cog is an aggregate for several cognitive tests intended to provide a global cognitive score and consists of 11 tasks. The tasks (and corresponding score range)) are Word Recall (0-10), Naming (0-4), Commands (0-5), Constructional Praxis (0-5) Ideational Praxis (0-5), Orientation (0-8), Word Recognition (0-12), Language (0-5), Word Finding Difficulty (0-5), and Remembering Test Instructions (1-5). The range of aggregate scores (sum of scores) is 1 to 69, with higher scores meaning worse cognitive performance. The change was calculated subtracting the baseline score from the final visit score.
Time Frame: 12 months
Population: Analyses used an intent to treat approach with last observation carried forward
Measure: Mean (Standard Deviation); unit: score
Groups:
- Placebo: placebo identical to metformin.
  placebo: placebo identical to metformin 2 tablets twice a day titrated from one table once a day. Participants were maintained on the highest tolerated dose (0,1,2,3,4 tablets).
- Metformin: metformin 1000 mg twice a day
  metformin: metformin 1000 mg twice a day titrated from 500 mg once a day.Participants were maintained on the highest tolerated dose (0,1,2,3,4 tablets of 500 mg each).
Arm/Group | Placebo | Metformin
Number analyzed (Participants) | 40 | 40
score | -1.98 (5.5) | 0.0 (3.3)
Statistical Analysis 1: Comparison: Placebo vs Metformin; Test type: Superiority or Other; p = 0.06, t-test, 2 sided; Mean Difference (Final Values) = 1.98, Standard Deviation 1.01 — The difference is the value for the metformin arm minus the value for the placebo arm
Statistical Analysis 2: Comparison: Placebo vs Metformin; Test type: Superiority or Other; p = 0.34, ANCOVA; adjusted for baseline ADAS-Cog score; Mean Difference (Final Values) = 0.9, Standard Deviation 0.91 — The difference is the value for the metformin arm minus the value for the placebo arm

3. Secondary Outcome: Change in Relative Glucose Uptake (rCMRg) in the Posterior Cingulate-precuneus.
Description: Change in relative glucose uptake (rCMRgl) in the posterior cingulate-precuneus measured with subscale (ADAS-Cog) from brain [18]F-labeled 2-deoxy-2-fluoro-D-glucose (FDG) positron emission tomography (PET). The unit for rCMRgl is %. The results presented are absolute differences in rCMRgl, presented in % units; the change was calculated subtracting the baseline rCMRgl from the follow-up rCMRgl
Time Frame: 12 months
Population: Out of 40 persons recruited in the imaging sub study, 33 underwent a 12 month scan (18 in the placebo group, 15 in the metformin group).
Measure: Mean (Standard Deviation); unit: percentage of rCMRgl
Groups:
- Placebo: Placebo identical to metformin.
  placebo: placebo identical to metformin 2 tablets twice a day titrated from one table once a day. Participants remained on the highest tolerated dose (0,1,2,3,4 tablets).
Arm/Group | Placebo | Metformin
Number analyzed (Participants) | 18 | 15
percentage of rCMRgl | 0.0 (6.0) | 2.0 (6.3)
Statistical Analysis 1: Comparison: Placebo vs Metformin; Test type: Superiority or Other; p = 0.36, t-test, 2 sided; Mean Difference (Final Values) = 2.0, Standard Deviation 2.14 — The difference is the value for the metformin arm minus the value for the placebo arm

4. Other Pre Specified Outcome: Change in Plasma Amyloid Beta-42
Description: Change in plasma Amyloid beta-42 from baseline to 12 months
Time Frame: 12 months
Measure: Mean (Standard Deviation); unit: pg/ml
Groups:
- Metformin: metformin 1000 mg twice a day
  metformin: metformin 1000 mg twice a day titrated from 500 mg once a day.Participants remained on the highest tolerated dose (0,1,2,3,4 tablets of 500 mg each).
Arm/Group | Placebo | Metformin
Number analyzed (Participants) | 40 | 40
pg/ml | -4.40 (23.51) | 0.69 (18.5)
Statistical Analysis 1: Comparison: Placebo vs Metformin; Test type: Superiority or Other; p = 0.34, t-test, 2 sided; Mean Difference (Net) = 5.09, Standard Deviation 4.73 — The difference is the value for the metformin arm minus the value for the placebo arm

ADVERSE EVENTS:
Time Frame: 12 months
Description: The adverse event data were collected during the 12 months of the duration of the trial
Groups:
- Placebo: Matching placebo
  placebo: matching identical to metformin 2 tablets twice a day titrated from one table once a day
Arm/Group | Placebo | Metformin
Serious Adverse Events (participants affected / at risk) | 0/40 | 0/40
Other Adverse Events (participants affected / at risk) | 0/40 | 3/40
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=40) | Metformin (N=40)
Gastrointestinal symptoms (Gastrointestinal disorders) | 0 (0) | 3 (3)

LIMITATIONS AND CAVEATS:
The pilot study had a small sample size and relatively short duration, both for the whole sample, and the imaging sub-sample

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No